CLINICAL TRIAL: NCT03480828
Title: Diaphragm Ultrasound to Predict Weaning Outcomes in Mechanically Ventilated Patients
Status: Completed | Type: Observational
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of the anesthesia and intensive care department, Mongi Slim Hospital
Other Study IDs: rea1
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Accuracy of DE and DTF in Prediction of Extubation Success

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: comparaison between DE and DTF in prediction of extubation success — diaphragm ultrasound and measurement of DE and DTF in patients meeting all extubation criteria during spontaneous breathing trial

SUMMARY:
This trial enrolled all the adult patients who were mechanically ventilated for more than 48 hours and met all creteria for extubation. Patients who needed reintubation for upper aiway obstruction, neurological or hemodynamic alteration were excluded. The diaphragm ultrasound was performed during spontaneous breathing test or pressure support ventilation trial measuring the dipahragmatic excursion (DE) and the diaphragm thickening fraction (DTF) whithin 24 hours before extubation.

DETAILED DESCRIPTION:
This trial enrolled all the adult patients who were mechanically ventilated for more than 48 hours and met all creteria for extubation. Patients who needed reintubation for upper aiway obstruction, neurological or hemodynamic alteration were excluded. The diaphragm ultrasound was performed during spontaneous breathing test or pressure support ventilation trial measuring the dipahragmatic excursion (DE) and the diaphragm thickening fraction (DTF) whithin 24 hours before extubation. The investigators compared the median values of DE and DTF in the group of successfully extubated patients and the group of patients who needed reintubation.

Our study compared the utility of DTF and DE to predict extubation success.

ELIGIBILITY:
Inclusion Criteria:

* patients who were mechanically ventilated for more than 48h and meeting all criteria for extubation
* patients without history of neuromuscular disease, or severe chronic respiratory failure

Exclusion Criteria:

* patients who needed reintubation for upper airway obstruction or neurological or hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who were mechanically ventilated for more than 48 hours and meeting all extubation criteria without a history of neuromuscular disease or severe chronic respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
extubation success | 48 hours after extubation
  comparaison between DE and DTF values in successfully extubated patients

CONTACTS AND LOCATIONS:
Overall Officials: Mhamed Sami Mebazaa, Professor, Principal Investigator — Mongi Slim Hospital
Locations (1):
- Mongi Slim Hospital, La Marsa, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided